CLINICAL TRIAL: NCT00005209
Title: Genetic Epidemiology of Coronary Heart Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1088; R01HL039107 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2008-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease

SUMMARY:
To relate observations at the DNA level to the distribution of coronary heart disease in the population at large.

DETAILED DESCRIPTION:
BACKGROUND:

The Rochester Family Heart Study was initiated in 1983 to study the genetic basis for familial aggregation of apolipoprotein A-I and hypertension in Rochester, Minnesota. Recruitment began in 1985 and resulted in data on 2,259 individuals in 300 three generation pedigrees. The study was supported by R01HL24489.

Lipid levels play a central role in determining the predisposition to coronary heart disease. In Western industrialized societies diseases of the heart rank as the number one cause of morbidity and mortality in the adult population. Thirty percent of all deaths in the United States in 1982 were attributable to coronary heart disease. Epidemiological studies of total communities including Framingham, Massachusetts and Tecumseh, Michigan have established a long list of factors that predict increased risk to coronary heart disease. Those that have been implicated include male gender, aging, positive family history, sedentary life style, diabetes, high blood pressure, cigarette smoking, overweight and abnormal plasma levels of lipids and lipoproteins. Although there is great variation among individuals in the risk factors associated with the development of coronary heart disease, the disease typically involves the infiltration of cholesterol into the intimal wall of the arteries beginning early in life. It has been hypothesized that each individual inherits or experiences an array of risk factors that determine susceptibility to the disease process that progresses through the phases of injury to the vascular wall, infiltration of lipids, accumulation of cholesterol esters, a proliferation of cells, stenosis and finally occlusion that leads to the coronary heart disease outcome. Lipid metabolism plays a central role in determining the progression of this process. A role for elevated lipids in the etiology of coronary heart disease is supported by the Lipid Research Clinics trial of cholestyramine which established that a 20 percent reduction of plasma low density lipoprotein (LDL) in particular, results in a 19 percent reduction of coronary heart disease after seven years in high risk males. Most studies to date have focused on environmental factors associated with variability in risk factors. Biometrical studies have estimated the role of genes in determining interindividual variability in lipid and lipoprotein phenotypes by comparing and contrasting the levels in related and unrelated individuals living together and apart. With the advent of new techniques to measure variability in gene products and at the DNA level, it is now possible to expand our studies of the role of genes in both lipid metabolism and coronary heart disease. Knowledge about the genetic epidemiology of coronary heart disease will provide valuable tools for clinical screening and diagnosis and will make it possible to develop a rational strategy to intervene. Not all individuals respond in the same way to lipid-lowering strategies. By knowing the genes involved in regulating the metabolic factors that are altered in coronary heart disease we will be able to sort out those individuals who will respond to specific treatments.

DESIGN NARRATIVE:

Beginning in 1987 and using blood samples and data from the RFHS, variation at the DNA level was determined using restriction fragment length polymorphisms and at the protein level by isoelectric focusing. The relationships were defined in the population among the apolipoproteins, cholesterol, triglycerides, high density lipoprotein cholesterol phenotypes and estimates were done on the effects of age, sex, smoking, drug use, and obesity on these relationships. Estimates were determined for the fraction of interindividual variation in the apos attributable to gene loci coding for these molecules. Estimates were also determined for the fraction of interindividual variation in cholesterol, triglycerides, and high density lipoprotein cholesterol attributable to gene loci coding for the apos and the LDL receptor. A determination was also made as to whether genotypic variation for the gene loci coding for the apo and LDL-receptor contributed to the prediction of coronary heart disease beyond that provided by the effects of these gene loci on the interindividual variation in the apos, cholesterol, triglycerides, and high density lipoprotein cholesterol. Radioimmunoassay and medical information collection took place at the Mayo Clinic. DNA probes, DNA studies of special families, and definition of new restriction fragment length polymorphism took place at Charing Cross Hospital in London, England. RFLP typing of genes coding for the apolipoproteins and the LDL receptor and electrophoretic typing of the known apo E and AIV protein polymorphisms took place at the University of Pittsburgh. The genetic architecture responsible for phenotypic variability in the population at large was defined at the University of Michigan and Washington University, St. Louis.

The study was renewed in 1992 to carry out six aims that 1) provided new information about four polymorphic genes involved in reverse cholesterol transport; 2) completed the investigators' studies to evaluate the utility of genetic variation in 12 candidate genes for prediction of coronary artery disease; 3) identified individuals who carry mutations that have an impact on coronary artery disease; and 4) began molecular studies of these individuals to define the DNA changes that are responsible. New noninvasive measures of coronary artery disease in asymptomatic individuals using ultrafast cardiac computed tomography complemented efforts to evaluate the role of measured genetic variation in predicting coronary artery disease.

The study was renewed again in 1997 with five specific aims. Aims 1 and 2 identified genomic regions containing new coronary artery disease susceptibility genes, using 234 tandem repeat marker loci at a 10 centimorgan (cM) density and the variance component method of linkage in 274 multigeneration pedigrees, both globally and in particular contexts defined by gender, age, body mass index and smoking. For those regions that showed linkage, confirmatory linkage analysis was conducted in a second independent sample of 301 multigeneration pedigrees. In regions where linkage was replicated, fine structure linkage analyses was conducted, using additional marker loci, located approximately every 1 cM. Specific aims 3 and 4 identified functional DNA variations in the new candidate coronary artery disease susceptibility genes. Direct DNA sequencing and cladistic analyses were used to estimate the average, context dependent, dominant, and epistatic effects associated with these functional DNA variations. Specific aim 5 estimated the association between the risk of coronary artery disease and functional genotypes identified by the cladistic analyses carried out in specific aims 3 and 4 before and after considering the intermediate biological risk factors that link the effects of genetic and environmental variation to variation in risk of disease.

The study was renewed in 2001 through July 2006 to continue to investigate innovative analytic and molecular aspects of risk of coronary artery disease, in particular, the contribution of polymorphic variation at the ApoE locus and two other candidate regions of the genome on variation in plasma ApoE level.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1987-08; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Sing — University of Michigan

REFERENCES:
- [Background] Pairitz G, Davignon J, Mailloux H, Sing CF. Sources of interindividual variation in the quantitative levels of apolipoprotein B in pedigrees ascertained through a lipid clinic. Am J Hum Genet. 1988 Sep;43(3):311-21. PMID 3414686
- [Background] Davignon J, Gregg RE, Sing CF. Apolipoprotein E polymorphism and atherosclerosis. Arteriosclerosis. 1988 Jan-Feb;8(1):1-21. doi: 10.1161/01.atv.8.1.1. PMID 3277611
- [Background] Templeton AR, Sing CF, Kessling A, Humphries S. A cladistic analysis of phenotype associations with haplotypes inferred from restriction endonuclease mapping. II. The analysis of natural populations. Genetics. 1988 Dec;120(4):1145-54. doi: 10.1093/genetics/120.4.1145. PMID 3147219
- [Background] Kaprio J, Ferrell RE, Kottke BA, Sing CF. Smoking and reverse cholesterol transport: evidence for gene-environment interaction. Clin Genet. 1989 Oct;36(4):266-8. doi: 10.1111/j.1399-0004.1989.tb03201.x. No abstract available. PMID 2509115
- [Background] Reilly SL, Kottke BA, Sing CF. The effects of generation and gender on the joint distributions of lipid and apolipoprotein phenotypes in the population at large. J Clin Epidemiol. 1990;43(9):921-40. doi: 10.1016/0895-4356(90)90076-2. PMID 2213081
- [Background] Kottke BA, Friedlaender JS, Zerba KE, Sing CF. Lipid and apolipoprotein levels in six Solomon Island societies differ from those in a U.S. white population. Am J Phys Anthropol. 1990 Apr;81(4):483-91. doi: 10.1002/ajpa.1330810405. PMID 2110417
- [Background] Sing CF, Haviland MB, Zerba KE, Templeton AR. Application of cladistics to the analysis of genotype-phenotype relationships. Eur J Epidemiol. 1992 May;8 Suppl 1:3-9. doi: 10.1007/BF00145343. PMID 1354623
- [Background] Sing CF, Haviland MB, Templeton AR, Zerba KE, Reilly SL. Biological complexity and strategies for finding DNA variations responsible for inter-individual variation in risk of a common chronic disease, coronary artery disease. Ann Med. 1992 Dec;24(6):539-47. doi: 10.3109/07853899209167008. PMID 1485951
- [Background] Reilly SL, Ferrell RE, Kottke BA, Sing CF. The gender-specific apolipoprotein E genotype influence on the distribution of plasma lipids and apolipoproteins in the population of Rochester, Minnesota. II. Regression relationships with concomitants. Am J Hum Genet. 1992 Dec;51(6):1311-24. PMID 1463013
- [Background] Haviland MB, Kessling AM, Davignon J, Sing CF. Estimation of Hardy-Weinberg and pairwise disequilibrium in the apolipoprotein AI-CIII-AIV gene cluster. Am J Hum Genet. 1991 Aug;49(2):350-65. PMID 1678249
- [Background] Reilly SL, Ferrell RE, Kottke BA, Kamboh MI, Sing CF. The gender-specific apolipoprotein E genotype influence on the distribution of lipids and apolipoproteins in the population of Rochester, MN. I. Pleiotropic effects on means and variances. Am J Hum Genet. 1991 Dec;49(6):1155-66. PMID 1842218
- [Background] Kamboh MI, Ferrell RE, Kottke BA. Expressed hypervariable polymorphism of apolipoprotein (a). Am J Hum Genet. 1991 Nov;49(5):1063-74. PMID 1928089
- [Background] Crews DE, Kamboh MI, Bindon JR, Ferrell RE. Genetic studies of human apolipoproteins. XVII: Population genetics of apolipoprotein polymorphisms in American Samoa. Am J Phys Anthropol. 1991 Feb;84(2):165-70. doi: 10.1002/ajpa.1330840206. PMID 2021192
- [Background] Kamboh MI, Weiss KM, Ferrell RE. Genetic studies of human apolipoproteins. XVI. APOE polymorphism and cholesterol levels in the Mayans of the Yucatan Peninsula, Mexico. Clin Genet. 1991 Jan;39(1):26-32. doi: 10.1111/j.1399-0004.1991.tb02981.x. PMID 1997212
- [Background] Kamboh MI, Ferrell RE. Genetic studies of human apolipoproteins. XV. An overview of IEF immunoblotting methods to screen apolipoprotein polymorphisms. Hum Hered. 1990;40(4):193-207. doi: 10.1159/000153931. PMID 2199367
- [Background] Kwon JM, Boehnke M, Burns TL, Moll PP. Commingling and segregation analyses: comparison of results from a simulation study of a quantitative trait. Genet Epidemiol. 1990;7(1):57-68. doi: 10.1002/gepi.1370070113. PMID 2184092
- [Background] Ferrell RE, Kamboh MI, Majumder PP, Valdez R, Weiss KM. Genetic studies of human apolipoproteins. XIII. Quantitative polymorphism of apolipoprotein C-III in the Mayans of the Yucatan Peninsula. Hum Hered. 1990;40(3):127-35. doi: 10.1159/000153919. PMID 2365371
- [Background] Kamboh MI, Kelly LJ, Ferrell RE. Genetic studies of human apolipoproteins: XIV. A simple agarose isoelectric focusing gel method for apolipoprotein E phenotyping. Electrophoresis. 1990 Apr;11(4):314-8. doi: 10.1002/elps.1150110408. PMID 2340826
- [Background] Zerba KE, Friedlaender JS, Sing CF. Heterogeneity of the blood pressure distribution among Solomon Islands societies with increasing acculturation. Am J Phys Anthropol. 1990 Apr;81(4):493-511. doi: 10.1002/ajpa.1330810406. PMID 2333938
- [Background] Ferrell RE, Sepehrnia B, Kamboh MI, VandeBerg JL. Highly polymorphic apolipoprotein A-IV locus in the baboon. J Lipid Res. 1990 Jan;31(1):131-5. PMID 2313197
- [Background] Templeton AR, Crandall KA, Sing CF. A cladistic analysis of phenotypic associations with haplotypes inferred from restriction endonuclease mapping and DNA sequence data. III. Cladogram estimation. Genetics. 1992 Oct;132(2):619-33. doi: 10.1093/genetics/132.2.619. PMID 1385266
- [Background] Stengard JH, Zerba KE, Pekkanen J, Ehnholm C, Nissinen A, Sing CF. Apolipoprotein E polymorphism predicts death from coronary heart disease in a longitudinal study of elderly Finnish men. Circulation. 1995 Jan 15;91(2):265-9. doi: 10.1161/01.cir.91.2.265. PMID 7805227
- [Background] Reilly SL, Ferrell RE, Sing CF. The gender-specific apolipoprotein E genotype influence on the distribution of plasma lipids and apolipoproteins in the population of Rochester, MN. III. Correlations and covariances. Am J Hum Genet. 1994 Nov;55(5):1001-18. PMID 7977338
- [Background] Rastogi A, Bren ND, Hallaway BJ, Kottke BA. Immunomagnetic separation of subpopulations of apolipoprotein A-I. Mayo Clin Proc. 1994 Feb;69(2):137-43. doi: 10.1016/s0025-6196(12)61040-4. PMID 8309265
- [Background] Pettitt DJ, Moll PP, Knowler WC, Mott DM, Nelson RG, Saad MF, Bennett PH, Kottke BA. Insulinemia in children at low and high risk of NIDDM. Diabetes Care. 1993 Apr;16(4):608-15. doi: 10.2337/diacare.16.4.608. PMID 8462388
- [Background] Templeton AR, Sing CF. A cladistic analysis of phenotypic associations with haplotypes inferred from restriction endonuclease mapping. IV. Nested analyses with cladogram uncertainty and recombination. Genetics. 1993 Jun;134(2):659-69. doi: 10.1093/genetics/134.2.659. PMID 8100789
- [Background] Reilly SL, Sing CF, Savageau MA, Turner ST. Analysis of systems influencing renal hemodynamics and sodium excretion. I. Biochemical systems theory. Integr Physiol Behav Sci. 1994 Jan-Mar;29(1):55-73. doi: 10.1007/BF02691281. PMID 8018552
- [Background] Zerba KE, Ferrell RE, Sing CF. Genotype-environment interaction: apolipoprotein E (ApoE) gene effects and age as an index of time and spatial context in the human. Genetics. 1996 May;143(1):463-78. doi: 10.1093/genetics/143.1.463. PMID 8722796
- [Background] Haviland MB, Ferrell RE, Sing CF. Association between common alleles of the low-density lipoprotein receptor gene region and interindividual variation in plasma lipid and apolipoprotein levels in a population-based sample from Rochester, Minnesota. Hum Genet. 1997 Jan;99(1):108-14. doi: 10.1007/s004390050322. PMID 9003506
- [Background] Moore JH, Reilly SL, Ferrell RE, Sing CF. The role of the apolipoprotein E polymorphism in the prediction of coronary artery disease age of onset. Clin Genet. 1997 Jan;51(1):22-5. doi: 10.1111/j.1399-0004.1997.tb02408.x. PMID 9084929
- [Background] Stengard JH, Zerba KE, Turner ST, Sing CF. A biometrical study of the relationship between sodium-lithium countertransport and triglycerides. Ann Hum Genet. 1997 Mar;61(Pt 2):121-36. doi: 10.1046/j.1469-1809.1997.6120121.x. PMID 9177119
- [Background] Kardia SL, Sing CF, Turner ST. The response of renal plasma flow to angiotensin II infusion in a population-based sample and its association with the parental history of essential hypertension. J Hypertens. 1997 May;15(5):483-93. doi: 10.1097/00004872-199715050-00003. PMID 9170000
- [Background] Stengard JH, Pekkanen J, Sulkava R, Ehnholm C, Erkinjuntti T, Nissinen A. Apolipoprotein E polymorphism, Alzheimer's disease and vascular dementia among elderly Finnish men. Acta Neurol Scand. 1995 Oct;92(4):297-8. doi: 10.1111/j.1600-0404.1995.tb00132.x. PMID 8848934
- [Background] Kardia SL, Haviland MB, Sing CF. Correlates of family history of coronary artery disease in children. J Clin Epidemiol. 1998 Jun;51(6):473-86. doi: 10.1016/s0895-4356(98)00008-0. PMID 9635996
- [Background] Nelson MR, Kardia SL, Ferrell RE, Sing CF. Influence of apolipoprotein E genotype variation on the means, variances, and correlations of plasma lipids and apolipoproteins in children. Ann Hum Genet. 1999 Jul;63(Pt 4):311-28. doi: 10.1046/j.1469-1809.1999.6340311.x. PMID 10738543
- [Background] Schwartz GL, Turner ST, Moore JH, Sing CF. Predictors of interindividual variation in ambulatory blood pressure and their time or activity dependence. Am J Hypertens. 2000 Jan;13(1 Pt 1):52-60. doi: 10.1016/s0895-7061(99)00127-2. PMID 10678271
- [Background] Kardia SL, Haviland MB, Ferrell RE, Sing CF. The relationship between risk factor levels and presence of coronary artery calcification is dependent on apolipoprotein E genotype. Arterioscler Thromb Vasc Biol. 1999 Feb;19(2):427-35. doi: 10.1161/01.atv.19.2.427. PMID 9974428
- [Background] Zerba KE, Ferrell RE, Sing CF. Genetic structure of five susceptibility gene regions for coronary artery disease: disequilibria within and among regions. Hum Genet. 1998 Sep;103(3):346-54. doi: 10.1007/s004390050828. PMID 9799092
- [Background] Clark AG, Weiss KM, Nickerson DA, Taylor SL, Buchanan A, Stengard J, Salomaa V, Vartiainen E, Perola M, Boerwinkle E, Sing CF. Haplotype structure and population genetic inferences from nucleotide-sequence variation in human lipoprotein lipase. Am J Hum Genet. 1998 Aug;63(2):595-612. doi: 10.1086/301977. PMID 9683608
- [Background] Templeton AR, Weiss KM, Nickerson DA, Boerwinkle E, Sing CF. Cladistic structure within the human Lipoprotein lipase gene and its implications for phenotypic association studies. Genetics. 2000 Nov;156(3):1259-75. doi: 10.1093/genetics/156.3.1259. PMID 11063700
- [Background] Fullerton SM, Clark AG, Weiss KM, Nickerson DA, Taylor SL, Stengard JH, Salomaa V, Vartiainen E, Perola M, Boerwinkle E, Sing CF. Apolipoprotein E variation at the sequence haplotype level: implications for the origin and maintenance of a major human polymorphism. Am J Hum Genet. 2000 Oct;67(4):881-900. doi: 10.1086/303070. Epub 2000 Sep 13. PMID 10986041
- [Background] Nelson MR, Kardia SL, Ferrell RE, Sing CF. A combinatorial partitioning method to identify multilocus genotypic partitions that predict quantitative trait variation. Genome Res. 2001 Mar;11(3):458-70. doi: 10.1101/gr.172901. PMID 11230170
- [Background] Fullerton SM, Clark AG, Weiss KM, Taylor SL, Stengard JH, Salomaa V, Boerwinkle E, Nickerson DA. Sequence polymorphism at the human apolipoprotein AII gene ( APOA2): unexpected deficit of variation in an African-American sample. Hum Genet. 2002 Jul;111(1):75-87. doi: 10.1007/s00439-002-0763-x. Epub 2002 Jun 14. PMID 12136239
- [Background] Wilund KR, Ferrell RE, Phares DA, Goldberg AP, Hagberg JM. Changes in high-density lipoprotein-cholesterol subfractions with exercise training may be dependent on cholesteryl ester transfer protein (CETP) genotype. Metabolism. 2002 Jun;51(6):774-8. doi: 10.1053/meta.2002.32730. PMID 12037734
- [Background] Hagberg JM, Zmuda JM, McCole SD, Rodgers KS, Ferrell RE, Wilund KR, Moore GE. Moderate physical activity is associated with higher bone mineral density in postmenopausal women. J Am Geriatr Soc. 2001 Nov;49(11):1411-7. doi: 10.1046/j.1532-5415.2001.4911231.x. PMID 11890577
- [Background] Stengard JH, Clark AG, Weiss KM, Kardia S, Nickerson DA, Salomaa V, Ehnholm C, Boerwinkle E, Sing CF. Contributions of 18 additional DNA sequence variations in the gene encoding apolipoprotein E to explaining variation in quantitative measures of lipid metabolism. Am J Hum Genet. 2002 Sep;71(3):501-17. doi: 10.1086/342217. Epub 2002 Aug 5. PMID 12165926
- [Background] Sing CF, Stengard JH, Kardia SL. Genes, environment, and cardiovascular disease. Arterioscler Thromb Vasc Biol. 2003 Jul 1;23(7):1190-6. doi: 10.1161/01.ATV.0000075081.51227.86. Epub 2003 May 1. PMID 12730090
- [Background] Fullerton SM, Buchanan AV, Sonpar VA, Taylor SL, Smith JD, Carlson CS, Salomaa V, Stengard JH, Boerwinkle E, Clark AG, Nickerson DA, Weiss KM. The effects of scale: variation in the APOA1/C3/A4/A5 gene cluster. Hum Genet. 2004 Jun;115(1):36-56. doi: 10.1007/s00439-004-1106-x. Epub 2004 Apr 24. PMID 15108119
- [Background] Klos KL, Kardia SL, Hixson JE, Turner ST, Hanis C, Boerwinkle E, Sing CF. Linkage analysis of plasma ApoE in three ethnic groups: multiple genes with context-dependent effects. Ann Hum Genet. 2005 Mar;69(Pt 2):157-67. doi: 10.1046/j.1529-8817.2004.00148.x. PMID 15720297
- [Background] Klos KL, Hamon S, Clark AG, Boerwinkle E, Liu K, Sing CF. APOA5 polymorphisms influence plasma triglycerides in young, healthy African Americans and whites of the CARDIA Study. J Lipid Res. 2005 Mar;46(3):564-71. doi: 10.1194/jlr.M400437-JLR200. Epub 2004 Dec 16. PMID 15604515
- [Background] Kardia SL, Turner ST, Schwartz GL, Moore JH. Linear dynamic features of ambulatory blood pressure in a population-based study. Blood Press Monit. 2004 Oct;9(5):259-67. doi: 10.1097/00126097-200410000-00006. PMID 15472499
- [Background] Templeton AR, Maxwell T, Posada D, Stengard JH, Boerwinkle E, Sing CF. Tree scanning: a method for using haplotype trees in phenotype/genotype association studies. Genetics. 2005 Jan;169(1):441-53. doi: 10.1534/genetics.104.030080. Epub 2004 Sep 15. PMID 15371364
- [Background] Neel JV, Julius S, Weder A, Yamada M, Kardia SL, Haviland MB. Syndrome X: is it for real? Genet Epidemiol. 1998;15(1):19-32. doi: 10.1002/(SICI)1098-2272(1998)15:13.0.CO;2-#. PMID 9523208
- [Background] Sing CF, Moll PP. Genetics of atherosclerosis. Annu Rev Genet. 1990;24:171-87. doi: 10.1146/annurev.ge.24.120190.001131. No abstract available. PMID 2088166